CLINICAL TRIAL: NCT05539170
Title: Parents' Differential Susceptibility to a Randomized Controlled Microtrial: The Role of Physiological Signals as Underlying Mechanism
Brief Title: Parents' Differential Susceptibility to Microtrial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tilburg University (Other)
Responsible Party: Principal Investigator, Rabia Chhangur, Assistant professor, Tilburg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: TSB_RP604
Record Dates: First submitted 2022-09-06; First posted 2022-09-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-04

CONDITIONS: Parenting; Child Behavior; Parent-Child Relations
Keywords: differential susceptibility; parenting; intervention efficacy; randomized controlled microtrial
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Intervention Model Description: "micro" parenting intervention vs. care-as-usual control condition
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- "micro" parenting intervention (Experimental): Parents will be instructed to bring the completed questionnaires with them to the university lab. Then, in the lab, parents will be observed interacting with their child. Following these baseline conditions, half of the parents will receive the "micro" parenting intervention-in the form of individual positive feedback concerning their parenting and their child's behavior.
  Interventions: Behavioral: Immediate positive parenting feedback
- care-as-usual condition (No Intervention): Participants in the care-as-usual control condition receive no immediate positive parenting feedback but will also be taken aside without their child, receiving only the instructions of the experiment.

INTERVENTIONS:
Behavioral: Immediate positive parenting feedback — Individual positive feedback concerning their parenting and their child's behavior.
  Arms: "micro" parenting intervention

SUMMARY:
This randomized controlled microtrial, not just focus on parental (and child) responsiveness but also on an underlying physiological mechanism hypothesized to contribute to heightened susceptibility to parenting interventions.

DETAILED DESCRIPTION:
After being informed about the study, all participants giving written informed consent will be randomly assigned to the "micro" intervention condition (i.e., immediate positive parenting feedback) or care-as-usual control condition in a singe-blind manner in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Parents with children aged 4-6 years.

Exclusion Criteria:

* psychiatric/neurological disorder (as reported by the parent)
* mental retardation (IQ < 70)
* not mastering the Dutch language, and
* that their child is not living in another household during the weekdays

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Parental self-efficacy beliefs assessed with the General Scale of Parental Self-Efficacy Beliefs (GSPSEB) at pretest, posttest and follow-up | Parenting change: baseline (pretest), after 2 weeks (posttest), and after 4 weeks (follow-up)
  This 25-item scale is related to five domain-specific SEB factors: Discipline, Nurturance, Playing, Instrumental Care, and Teaching. Self-efficacy beliefs in parenting can be evaluated as a quantitative construct by asking parents their beliefs in specific parenting activities, such as teaching, playing, providing instrumental care, nurturing or disciplining their child. Items are in the form of affirmatives, for example: ''I am able to sense when my child is starting to become distressed'' for the Nurturance subscale. The items will be rated on a 5-point scale (1 = strongly disagree to 5 = strongly agree).
Parenting behavior assessed with the short version of the Parental Behavior Scale (PBS-S) at pretest, posttest and follow-up | Parenting change: baseline (pretest), after 2 weeks (posttest), and after 4 weeks (follow-up)
  This questionnaire consists of 25 items and comprises five subscales: Positive parenting (e.g., "I make time to listen to my child, when he/she wants to tell me something"), Discipline (e.g., "When my child has been disobedient, I give him/her a chore as punishment"), Harsh Punishment (e.g., "I spank my child when he/she is disobedient or naughty"), Material Rewarding (e.g., "I give my child candy as a reward for good behavior"), and Rule Setting (e.g., "I teach my child to be polite at school"). A 5-point scale is provided for each item, ranging from 1 = (almost) never to 5 = (almost) always.
Observed parenting behavior assessed with the Crowell Parent-Child interaction taks at pretest and posttest | Parenting change: baseline/pretest observation at lab (before intervention) and posttest observation at same labvisit (after intervention)
  The Crowell observation task takes 20 minutes to complete and consists of four episodes: warm-up, free play, frustration task, and recovery time. The parent scales (i.e., positive affect, autonomy support, negative affect, withdrawal, controlling behavior and laxness/inconsistent) are each internally consistent and well-defined conceptually. High internal consistency for each scale provides support for the reliability of the rating scale, and suggests that the Crowell scores can be useful as scale to measure caregiver responsiveness, but also collectively as a total score assessing overall relational functioning.

SECONDARY OUTCOMES:
Child externalizing problem assessed with the Eyberg Child Behavior Inventory (ECBI) at pretest, posttest and follow-up. | Change in child behavior: baseline (pretest), after 2 weeks (posttest), and after 4 weeks (follow-up)
  One subscale assessing the degree to which child externalizing problem is a problem from the 36-item Eyberg Child Behavior Inventory (ECBI) will be used to assess the occurrence of child externalizing problem behavior. This "Intensity" subscale measures frequency of externalizing behavior in children aged 2 to 16 years and has been shown to be a reliable (screening) instrument (3). Example items are: "Does not obey house rules" and "Whines."
Observed child behavior assessed with the Crowell Parent-Child interaction taks at pretest and posttest | Change in child behavior: baseline/pretest observation at lab (before intervention) and posttest observation at same labvisit (after intervention)
  The Crowell observation task takes 20 minutes to complete and consists of four episodes: warm-up, free play, frustration task, and recovery time. The child scales (i.e., positive affect, persistence/enthusiasms, irritability/negative affect, and noncompliance) are each internally consistent and well-defined conceptually. High internal consistency for each scale provides support for the reliability of the rating scale, and suggests that the Crowell scores can be useful as scale to measure child's affective presentation, but also collectively as a total score assessing overall relational functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Rabia R. Chhangur, PhD, Principal Investigator — Tilburg University
Locations (1):
- Tilburg School of Social and Behavioral Sciences, Tilburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chhangur RR, Belsky J. Parents' differential susceptibility to a "micro" parenting intervention: Rationale and study protocol for a randomized controlled microtrial. PLoS One. 2023 Mar 22;18(3):e0282207. doi: 10.1371/journal.pone.0282207. eCollection 2023. PMID 36947489